CLINICAL TRIAL: NCT01196351
Title: Effect of Activity at the Ventilation Threshold on Appetite and Food Intake After a Glucose Drink in Normal Weight, Overweight and Obese Boys
Brief Title: Activity at Ventilation Threshold on Appetite and Food Intake in Boys
Acronym: VeT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: G. Harvey Anderson, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CIHR-Kids21595_EXR1; CIHR (Other Grant/Funding Number: 482209)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Obesity Prevention
Keywords: boys; obesity; physical activity; exercise
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sedentary activity, noncaloric beverage (Experimental)
  Interventions: Other: Dietary Supplement: water with noncalorie sweetener
- Sedentary activity, glucose beverage (Experimental)
  Interventions: Other: Dietary Supplement: water with noncalorie sweetener
- Exercise activity, noncaloric beverage (Experimental)
  Interventions: Other: Activity: With noncalorie sweetener or glucose
- Exercise activity, glucose beverage (Experimental)
  Interventions: Other: Activity: With noncalorie sweetener or glucose

INTERVENTIONS:
Other: Dietary Supplement: water with noncalorie sweetener
  Arms: Sedentary activity, glucose beverage; Sedentary activity, noncaloric beverage
Other: Activity: With noncalorie sweetener or glucose
  Arms: Exercise activity, glucose beverage; Exercise activity, noncaloric beverage

SUMMARY:
The investigators hypothesize exercise increases short term appetite and food intake, and interferes with satiety and satiations to a preload in normal weight, overweight and obese boys.

DETAILED DESCRIPTION:
The effect of exercise (EXR) on short-term food intake (FI) and subjective appetite was investigated in normal weight (NW), overweight (OW) and obese (OB) boys were randomized into 4 treatments. Each boy consumed either a non-caloric sweetened control (CON) or GLU drink after either exercise (EXR) or sedentary activity. Subjects exercised at their ventilation threshold (VeT).

ELIGIBILITY:
Inclusion Criteria:

* Healthy boys with no emotional, behavioral or learning problems

Exclusion Criteria:

* Girls

Ages: 9 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
food intake (kcal) | at 30-35 min after the treatment

SECONDARY OUTCOMES:
Subjective appetite | 0-80 min

CONTACTS AND LOCATIONS:
Overall Officials: Harvey G. Anderson, PhD., Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bellissimo N, Desantadina MV, Pencharz PB, Berall GB, Thomas SG, Anderson GH. A comparison of short-term appetite and energy intakes in normal weight and obese boys following glucose and whey-protein drinks. Int J Obes (Lond). 2008 Feb;32(2):362-71. doi: 10.1038/sj.ijo.0803709. Epub 2007 Aug 14. PMID 17700578
- [Background] Bellissimo N, Thomas SG, Goode RC, Anderson GH. Effect of short-duration physical activity and ventilation threshold on subjective appetite and short-term energy intake in boys. Appetite. 2007 Nov;49(3):644-51. doi: 10.1016/j.appet.2007.04.004. Epub 2007 Apr 22. PMID 17537539
- [Background] Bozinovski NC, Bellissimo N, Thomas SG, Pencharz PB, Goode RC, Anderson GH. The effect of duration of exercise at the ventilation threshold on subjective appetite and short-term food intake in 9 to 14 year old boys and girls. Int J Behav Nutr Phys Act. 2009 Oct 9;6:66. doi: 10.1186/1479-5868-6-66. PMID 19818131